CLINICAL TRIAL: NCT02778282
Title: MySafeRx™: An Integrated Mobile Platform for Buprenorphine Adherence
Acronym: MySafeRx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Zev Schuman-Olivier, Instructor, Departments of Psychiatry and Biomedical Data Sciences, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA040086 D14047; 1R34DA040086 (NIH)
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard Care through office-based opioid treatment with buprenorphine/naloxone and weekly urine toxicology screening
- Standard Care + MySafeRx™ Intervention (Experimental): The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing. This arm represents Standard Care plus MySafeRx™.
  Interventions: Other: MySafeRx™

INTERVENTIONS:
Other: MySafeRx™ — The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing.
  Arms: Standard Care + MySafeRx™ Intervention

SUMMARY:
The goal of the MySafeRx study is to evaluate the feasibility, acceptability, and usability of a novel platform that integrates text messaging reminders, secure electronic pill organizers, and daily remote brief motivational recovery support visits with a standardized protocol for supervised self- administration of buprenorphine via videoconferencing.

DETAILED DESCRIPTION:
Opioid use disorder is a serious public health issue. Buprenorphine/ Naloxone (B/N) is a partial opioid mu-receptor agonist dosed daily that prevents opioid withdrawal, blocks opioid euphoria and can prevent opioid overdose. Extended treatment with B/N increases rates of abstinence and outpatient treatment retention and decreases Hepatitis C (HCV) transmission. B/N treatment dropout is associated with relapse and overdose death.

B/N adherence may be a critical factor influencing retention and reducing overall healthcare costs. Also, B/N diversion is associated with poor adherence and has become increasingly common and worrisome. While many patients achieve stability after starting B/N treatment, more than 80% of 18-25 year olds leave treatment within a year with relapse as the most common reason. Ongoing illicit opioid use during treatment increases odds of relapse and dropout. The MySafeRx™ platform helps prescribers offer a higher level of support for vulnerable patients with opioid use disorder during periods of clinical instability. The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of B/N medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing. By offering this recovery support and medication adherence monitoring program during periods of instability, this system could improve treatment outcomes by ensuring increased adherence, while also preventing B/N diversion.

This study primarily seeks to demonstrate the feasibility, acceptability, and usability of the MySafeRx™ platform among young adults (18-39 years, inclusive) with opioid use disorders. While each key component may have an individual therapeutic effect, we hypothesize that an integrated process involving all key components may be necessary to unlock the full therapeutic potential of a mobile platform for daily remote supervised self-administration and diversion prevention among this group. Providing targeted motivational interviewing and recovery support at this context-specific moment of daily medication-taking when people are very receptive to treatment may offer a new opportunity for expanding how recovery support can be delivered. Usability will be assessed with the validated system usability scale as a primary outcome. Feasibility, acceptability and initial efficacy based on opioid urine toxicology will all be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men age 18-39, inclusive, who are competent, wish to participate and willing to provide informed consent.
2. DSM-V diagnosis of opioid use disorder, moderate or severe
3. Seeking to initiate buprenorphine treatment or currently receiving buprenorphine treatment but had recent positive illicit opioid urine toxicology or missed scheduled urine toxicology.

Exclusion Criteria:

1. DSM-V diagnosis of dementia, neurodegenerative disease, or other organic mental disorder, mental retardation, or autism.
2. Substantial cognitive impairment (Montreal Cognitive Assessment < 25/30)
3. Currently homeless
4. Actively homicidal or suicidal with an imminent plan
5. Serious unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease such that hospitalization for treatment of that illness is likely within the next 3 months.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with adequate medication adherence | Day 42
  Feasibility will be demonstrated by MySafeRx achieving supervised self-administration of B/N on >= 30 out of the first 42 days (equivalent to an average of 5 out of 7 days) for at least 2/3 of subjects randomized to MySafeRx.

SECONDARY OUTCOMES:
Acceptability | Day 42
  Level of patient acceptability (mean score > 3 out of 5 on the 13-item satisfaction scale)
Usability | 42 days
  Reported patient usability (mean score > 68 on the system usability scale)
Initial Clinical Efficacy-Illicit opioid use | 6 weeks
  Percent negative weekly opioid urine toxicology
Initial Clinical Efficacy-Medication adherence | 6 weeks
  Weekly self-reports of B/N adherence

OTHER OUTCOMES:
Treatment Retention | 6 weeks
  Percentage of patients dropped out from treatment or referred to higher level of care
Crisis and Hardship in Administering Office-Based Opioid Treatment (OBOT) Scale | 8 weeks
  Monthly CHAOS scale scores
Cost effectiveness ratio | 3 months
  Assess cost effectiveness ratio for prescribers and patients from MySafeRx™ versus standard care, which is the following [CE Ratio = (Cost{new}-Cost{current}) /(Effect{new}-Effect{current})

CONTACTS AND LOCATIONS:
Overall Officials: Zev D Schuman-Olivier, MD, Principal Investigator — Dartmouth College
Locations (3):
- United States (3):
  - Cambridge Health Alliance Outpatient Addiction Services, Somerville, Massachusetts
  - Hawthorn Recovery Center, Bennington, Vermont
  - Mount Anthony Primary Care, Bennington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schuman-Olivier Z, Weiss RD, Hoeppner BB, Borodovsky J, Albanese MJ. Emerging adult age status predicts poor buprenorphine treatment retention. J Subst Abuse Treat. 2014 Sep;47(3):202-12. doi: 10.1016/j.jsat.2014.04.006. Epub 2014 May 20. PMID 24953168
- [Background] Aaron Bangor, Philip T. Kortum & James T. Miller (2008) An Empirical Evaluation of the System Usability Scale, International Journal of Human-Computer Interaction, 24:6, 574-594, DOI: 10.1080/10447310802205776
- [Background] Schuman-Olivier Z, Borodovsky JT, Steinkamp J, Munir Q, Butler K, Greene MA, Goldblatt J, Xie HY, Marsch LA. MySafeRx: a mobile technology platform integrating motivational coaching, adherence monitoring, and electronic pill dispensing for enhancing buprenorphine/naloxone adherence during opioid use disorder treatment: a pilot study. Addict Sci Clin Pract. 2018 Sep 24;13(1):21. doi: 10.1186/s13722-018-0122-4. PMID 30249279
- See also: Website for Center for Technology and Behavioral Health at Dartmouth — http://www.c4tbh.org